CLINICAL TRIAL: NCT05772013
Title: Optimising Azithromycin Prevention Treatment in COPD to Reduce Exacerbations (OPACE): A Double Blind Adaptive Design Pragmatic Phase IV Randomised Controlled Trial
Brief Title: Optimising Azithromycin Prevention Treatment in COPD to Reduce Exacerbations
Acronym: OPACE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dr Ian B Wilkinson (Other)
Collaborators: University of Aberdeen (Other); NHS Greater Glasgow and Clyde (Other); University of East Anglia (Other); Nottingham City Hospital (Unknown); Swansea University (Other); Newcastle University (Other); University of Cambridge (Other); NHS Sunderland Clinical Commissioning Group (Unknown); Liverpool School of Tropical Medicine (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); University College London Hospitals (Other); Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Imperial College London (Other); Red Graphic (Unknown); Eramol (UK) Ltd. (Unknown); WGK Clinical Services Ltd. (Unknown); Sealed Envelope Ltd. (Unknown); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor-Investigator, Dr Ian B Wilkinson, Professor of Therapeutics, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCTU0333
Record Dates: First submitted 2023-02-27; First posted 2023-03-16 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Azithromycin; Chemoprophylaxis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: OPACE is a double-blind, adaptive design, placebo-controlled phase IV randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Continuous azithromycin (Active Comparator): Participants in this arm will continue with their standard of care (i.e. continuous dose of azithromycin according to their standard prescription) throughout the trial.
  Interventions: Drug: Azithromycin Pill
- Seasonal azithromycin (Other): Azithromycin will be taken by participants during the autumn-winter (October - March).
  Matched placebo will be taken by the participants in the spring-summer (April - September).
  Interventions: Drug: Azithromycin Pill; Drug: Placebo
- Complete Discontinuation of azithromycin (Placebo Comparator): Participants will take continuous matched placebo throughout the trial.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin Pill — Participants will take azithromycin according to their standard of care prescription.
  If the participant is on the seasonal azithromycin treatment arm, they will only take azithromycin during the winter months (October-March) followed by matched placebo (April-September).
  Arms: Continuous azithromycin; Seasonal azithromycin
Drug: Placebo — The placebo tablets will be matched in appearance, taste and smell to the azithromycin tablets.
  Arms: Complete Discontinuation of azithromycin; Seasonal azithromycin

SUMMARY:
People living with chronic obstructive pulmonary disease (COPD) may experience worsening of symptoms such as shortness of breath, cough and wheezing in addition to changes that may be expected for having COPD. The worsening of symptoms is called exacerbations or flare-ups and can be debilitating and frightening, requiring additional treatment, often with azithromycin. This is an antibiotic medicine that also has anti-inflammatory properties. It is prescribed as long-term prevention to reduce the risk of flare-ups. Some people may be affected by side effects from azithromycin. Antibiotic resistance is another concern, especially when using azithromycin for prevention rather than to treat active infection.

It is currently unclear as to whether people should be advised to stop taking azithromycin once COPD has stabilised, or to stop it over the summer when fewer flare-ups happen. It is also not known if azithromycin is more effective in some people or more likely to cause side effects in others. Given these uncertainties, it is challenging to know how best to use azithromycin in managing COPD. Azithromycin is a valuable antibiotic, and should be prescribed where it has benefit but avoid unnecessary side effects and reduce the chances of bacteria becoming resistant to it.

The purpose of this trial is to be able to gain results to answer these questions, and to establish the effects of stopping azithromycin in people whose COPD has stabilised, who have been taking it for at least 3 months. This trial will compare continuing azithromycin with stopping it completely, or stopping over the summer only, continuing over the winter. The investigators will compare the effects of these three treatments in the trial on flare-ups, symptoms and quality of life, and find out what factors may affect how individual participants respond to them.

DETAILED DESCRIPTION:
Background: Prophylactic azithromycin is recommended as a treatment to reduce the risk of chronic obstructive pulmonary disease (COPD) exacerbations in people with COPD at high risk of exacerbations. In clinical practice, there is much uncertainty in how to optimally use this valuable treatment in managing COPD. It is unknown whether azithromycin is effective beyond one-year of treatment; what happens when azithromycin is discontinued following a period of use; or temporarily discontinued over the summer when there are fewer exacerbations. Whether there are differences in treatment responsiveness between subgroups of people with COPD is also uncertain.

Aim: To evaluate the benefits and risks of complete or seasonal discontinuation of azithromycin chemoprophylaxis vs continued treatment in people with stable COPD at high risk of exacerbations and assess effects in participant subgroups.

Methods: Design: A randomised double-blinded, non-inferiority, adaptive-design pragmatic trial of 3 parallel arms (complete discontinuation, vs seasonal discontinuation vs continued azithromycin as standard of care), to test the strategy of discontinuation of prophylactic azithromycin in participants with stable COPD at high risk of exacerbations. Internal pilot to evaluate recruitment will run for 9 months from first participant first visit (FPFV).

Randomisation allocation will be 1:1:1. Adaptive design means a treatment arm can be dropped if futile at interim analysis, but remaining arms continue.

Setting: General Practitioner (GP) practices, specialist community clinics, hospitals.

Target population: Stable COPD participants prescribed azithromycin ≥3 months to reduce risk of COPD exacerbations.

Interventions assessed: Complete discontinuation of azithromycin (matched placebo), seasonal discontinuation (azithromycin October-March, matched placebo April-September), continued azithromycin (standard of care).

Trial duration and procedures: Median follow up will be 24 months. Participants will have up to 3 visits - baseline, 12 months, 24 months/end of trial, which may coincide with standard of care visits and be in-person or remote depending on participant's individual preference. Telephone follow-up will be conducted at 1 week, 3 months, 6 months, and 18 months. All participants will have active follow up until study end, even if primary endpoint met. If participants have 3 or more exacerbations/year they will be advised to stop their trial medication. Participants may restart regular azithromycin prescription after stopping trial medication if advised by their GP/specialist. Secondary outcomes will be collected over the entire trial period and therefore may include evaluation both on and off trial medication.

Outcome measures:

Primary endpoint: Time to first exacerbation (TTFE) necessitating additional treatment with antibiotics and/or corticosteroids.

Key secondary endpoints (collected over entire trial)

1. Number/rate and severity of exacerbations, length of exacerbation-free status
2. Health related quality of life measured by change in the EuroQol-5 dimension
3. Symptoms (COPD assessment tool (CAT) score and cough)
4. Side effects
5. Mortality
6. Cost effectiveness from National Health Service (NHS) perspective.

Sample size: 1311 participants (437 per arm). Assuming a median TTFE of 150 days and non-inferiority threshold of 30 days shorter, equates to the threshold on the hazard ratio scale of 1.25. Sample size is based on 90 percent power for two non-inferiority comparisons (seasonal and placebo compared with continuous as standard treatment), at 2.7 percent significance using a Cox proportional hazards model. Pre-specified factors for subgroup analysis include exacerbation history, forced expiratory volume at one second (FEV1 percentage) predicted, current/ex-smoking status, COPD Assessment Tool (CAT) score, age, blood eosinophils.

Conclusion:

This pragmatic, real world trial aims to answer the uncertainties regarding prophylactic azithromycin use in COPD.

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to provide informed consent.
* Have an established clinical diagnosis of COPD and be receiving prophylactic azithromycin for ≥ (at least) 3 months to reduce COPD exacerbations.
* Have a self-reported smoking history of ≥ (at least) 10 pack years.
* Be aged >= 40 years.
* Have clinically stable COPD, i.e. no COPD exacerbation for at least 6 weeks.

Exclusion Criteria:

* Known hypersensitivity to any of the trial drugs or excipients.
* Current breast feeding, pregnancy or planned pregnancy during the trial.
* Any medical history or clinically relevant abnormality that makes participant ineligible for inclusion because of a safety concern relating to continuing or discontinuing azithromycin or other considerations.
* Known immunodeficiency requiring immunoglobulin/specific antibody therapy.
* Azithromycin prophylaxis prescribed for non-COPD condition.
* Active participation in COPD Clinical Trial of an Investigational Medicinal Product (CTIMP).

Electrocardiograms (ECGs) will not be a trial assessment nor entry requirement.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1311 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
COPD exacerbation | Throughout the entire trial follow-up of 24 months
  Time to first COPD exacerbation.

SECONDARY OUTCOMES:
Number and rate of exacerbations | Throughout the entire trial follow-up of 24 months
  Number/rate of exacerbations (and differentiation by severity of exacerbations, i.e. requirement of hospitalisation)
Exacerbation-free period | Throughout the entire trial follow-up of 24 months
  Duration of exacerbation-free status
Treatment for respiratory indication | Throughout the entire trial follow-up of 24 months
  Antibiotics and/or corticosteroids use for respiratory indication
CAT Score | Throughout the entire trial follow-up of 24 months
  Symptoms/impact: COPD Assessment Tool (CAT) score
Cough visual analogue scale (VAS) score | Throughout the entire trial follow-up of 24 months
  The severity of the cough will be rated on a scale of 0 to 10, whereby 0 = no cough, 10 = worst cough
Health status | Throughout the entire trial follow-up of 24 months
  Measured by change in quality of life questionnaire: A scale of 0-100 will be used, whereby 0 = Worst health imaginable, 100 = Best health imaginable
Mortality | Throughout the entire trial follow-up of 24 months
  Mortality (all cause and specific)
Healthcare utilisation | Throughout the entire trial follow-up of 24 months
  Details about the number of hospitalizations and primary care consultations will be recorded. There will be linkage with NHS England and equivalent services.
Adverse events of special interest (AESI) and Serious Adverse Reactions (SARs) | Throughout the entire trial follow-up of 24 months
  AESI's include cardiovascular and hearing-defined as new prescription of hearing aids, liver function test (LFT) dysfunction). Serious adverse reactions (SARs) to be recorded as well.
Sputum culture results | Throughout the entire trial follow-up of 24 months
  Sputum culture results will only be obtained if clinically indicated and sample via routine clinical care to local lab. Record if positive result (i.e. name of organism cultured only, not cfu/ml). If multiple sent, most recent one to trial visit should be used.
Adherence to trial medication | Throughout the entire trial follow-up of 24 months
  Participants will be asked whether they have missed any doses of the trial medication, and if so, if they stopped taking it for longer than 2 weeks in duration and why. Participants will also be asked to return trial bottles and unused trial medication to the trial research team at their appointments.

CONTACTS AND LOCATIONS:
Overall Officials: Ian B Wilkinson, Study Director — University of Cambridge & University of Cambridge NHS Foundation Trust
Locations (1):
- Cambridge University Hospital NHS Trust, Addenbrookes Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR